CLINICAL TRIAL: NCT01370681
Title: An Open-label, Randomized, Crossover Study to Evaluate the Pharmacokinetics After Administration of CJ30001 and Co-administration of HKB0701/SLM0807 in Korean Healthy Subjects
Brief Title: A Pharmacokinetic Study of CJ30001 and HKB0701/SLM0807 in Healthy Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Geun Seog, Song / Director of Regulatory and Clinical Development, CJ Cheiljedang Corporation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_VCM_102
Record Dates: First submitted 2011-06-01; First posted 2011-06-10 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group1 (Experimental)
  Interventions: Drug: Period I : HKB0701 and SLM0807, Period II : CJ30001
- Group2 (Experimental)
  Interventions: Drug: Period I : CJ30001, Period II : HKB0701 and SLM0807

INTERVENTIONS:
Drug: Period I : HKB0701 and SLM0807, Period II : CJ30001
  Arms: Group1
Drug: Period I : CJ30001, Period II : HKB0701 and SLM0807
  Arms: Group2

SUMMARY:
The objective of this study is to demonstrate the bioequivalence of CJ30001(fixed-dose combination tablet of HKB0701 and SLM0807) relative to HKB0701 and SLM0807 co-administered to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who are in age range of 20-50years and the weight range is not exceed ±20% of ideal weight. Ideal weight = [height -100]*0.9
* Subjects with no history of any significant chronic disease
* Judged to be in good health on the basis of their vital sign, ECG, physical exam and routine laboratory data
* Available for the entire study period
* Willing to adhere to protocol requirements and sign a informed consent form

Exclusion Criteria:

* Subjects who have taken any drugs to induce or inhibit hepatic enzyme activity within 30days prior to drug administration
* Subjects who have symptom of an acute illness within 4 weeks prior to drug administration
* Subjects with a history of clinically significant allergies including drug allergies
* Subjects whose clinical laboratory test values are outside the accepted normal range(Especially,AST or ALT >1.25 times to normal range or total bilirubin > 1.5times to normal range)
* Subjects with a history of drug, caffeine abuse(caffeine drink >5cups/day)
* Subjects with a history of alcohol abuse(alcohol>30g/day) or who have ever drinked alcohol whinin 7days prior to drug administration
* Heavy smoker ( >10cigarettes/day)
* Subjects who have had a diet known to interfere with the absorption, distribution, metabolism or excretion of drugs (especially, consumption of grapefruit juice)
* Subjects who have donated plasma within 60days prior to drug administration
* Subjects who have participated in a clinical study within 90days prior to drug administration
* Subjects who have received any drugs that might confound the results of the trial in the opinion of principal investigator within 10days prior to drug administration (cimetidine within 7days prior to drug administration)
* Female subjects who are pregnant, breastfeeding or not using medically acceptable birth control

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Geometric mean Cmax | up to 24hrs
Geometric mean AUCt | up to 24hrs

CONTACTS AND LOCATIONS:
Overall Officials: Jae Gook Shin, MD, ph D, Principal Investigator — Inje University